CLINICAL TRIAL: NCT03898310
Title: UTI Prophylaxis With Cranberry Extract After Female Incontinence Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9977
Record Dates: First submitted 2019-02-27; First posted 2019-04-01 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Urinary Tract Infections; Incontinence
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry Extract Capsules (Experimental): 36mg of proanthocyanidins in cranberry capsules
  Interventions: Dietary Supplement: Cranberry extract capsules
- Placebo Capsules (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Cranberry extract capsules — Participants in the treatment arm will receive cranberry extract capsules.
  Arms: Cranberry Extract Capsules
Dietary Supplement: Placebo capsule — Participants in the placebo arm will receive placebo capsules.
  Arms: Placebo Capsules

SUMMARY:
The risk of urinary tract infection (UTI) following female incontinence surgery ranges between 6-48%. The literature has shown mixed results of the therapeutic efficacy of cranberry extract to prevent UTI in females, with some promising preliminary work in the prevention of UTI's following gynecologic surgery. The researchers will conduct a study of the effect of cranberry extracts on preventing urinary tract infections following mid urethral slings, which are the most common urinary incontinence procedures.

DETAILED DESCRIPTION:
The researchers are going to perform a randomized, double-blind, placebo controlled trial of cranberry extract capsules for the prevention of UTI following incontinence surgery. They will recruit patients from a single hospital in a 24 month duration. Eligible participants are women undergoing elective incontinence procedures that does not involve fistula repair or vaginal mesh excision. The therapeutic regimen will be Theracran One cranberry capsules containing 36mg of proanthocyanidins and placebo cranberry capsules and placebo capsules. Both will be supplied by Theralogix Nutritional Sciences.

Following randomization into treatment or placebo therapy, the participants will be asked to start prophylaxis on day of surgery for a duration of six weeks. The researchers will collect urine specimen via catheter upon insertion in the operating room. At time of discharge, the researchers will provide all participants with capsules for six weeks of the assigned regimen until they are seen for their post-operative visit.

Participants will be told to contact research staff immediately and collect a urine specimen should they experience urinary symptoms consistent with UTI. The researchers will administer a brief structured interview regarding type and duration of symptoms and refer for treatment when necessary. Urine will be cultured using standard microbiologic techniques for the presence of uropathogens at one clinical laboratory.

Participants will be asked to complete a self-administered questionnaire at the two week post-operative clinic visit and again at six weeks. At study exit, the researchers will collect capsule bottles to ensure and assess compliance.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective incontinence procedures that does not involve fistula repair or vaginal mesh excision

Exclusion Criteria:

* Women undergoing incontinence procedures involving fistula repair or vaginal mesh excision

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 141 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2023-01-22 (Actual); Study Completion 2023-01-22 (Actual)

PRIMARY OUTCOMES:
Urine culture based on type of symptoms | 2 weeks
  A urine culture to determine UTI will be performed based on symptoms such as urgency, frequency, dysuria or hematuria following incontinence surgery, as reported by the participant.

SECONDARY OUTCOMES:
Duration of symptoms | 2 weeks
  If symptoms are reported, the participant will be asked long they have had these symptoms since surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Lieschen Quiroz, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Temtanakitpaisan T, Buppasiri P, Lumbiganon P, Laopaiboon M, Rattanakanokchai S. Prophylactic antibiotics for preventing infection after continence surgery in women with stress urinary incontinence. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD012457. doi: 10.1002/14651858.CD012457.pub2. PMID 35349162